CLINICAL TRIAL: NCT00019747
Title: A Phase II Trial of Oral Thalidomide as an Adjuvant Agent Following Metastasectomy in Patients With Recurrent Colorectal Cancer
Brief Title: Surgery With or Without Thalidomide in Treating Patients With Recurrent or Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: DSMB recommended closure of the protocol due to slow accrual.
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, M.D., Dr. Steven Rosenberg, National Institutes of Health Clinical Center (CC)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 990102; 99-C-0102; CDR0000067098
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Results first posted 2012-10-25 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-09

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Thalidomide; Chemotherapy, Adjuvant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 - Thalidomide once daily (Experimental): Patients receive oral thalidomide 100 mg at bedtime once daily for 4 weeks, then progresses to 200 mg at bedtime for 4 weeks, then progresses to 300 mg at bedtime (maintenance dose).
  Interventions: Drug: thalidomide; Procedure: adjuvant therapy
- Arm 2 - Placebo once daily (Placebo Comparator): Patients receive oral placebo once daily.
  Interventions: Procedure: adjuvant therapy; Other: Placebo

INTERVENTIONS:
Drug: thalidomide — oral thalidomide 100 mg at bedtime once daily for 4 weeks, then progresses to 200 mg at bedtime for 4 weeks, then progresses to 300 mg at bedtime (maintenance dose).
  Other Names: Thalomid
  Arms: Arm 1 - Thalidomide once daily
Procedure: adjuvant therapy — Initial dose: 100 mg by mouth (po) every bedtime ( Q hs) for four weeks, then progress to 200 mg po Q hs for four weeks, then progress to maintenance dose: 300 mg po Q hs.
Other: Placebo — oral placebo once daily
  Arms: Arm 2 - Placebo once daily

SUMMARY:
RATIONALE: Thalidomide may stop the growth of colorectal cancer by stopping blood flow to the tumor. Giving thalidomide after surgery may kill any remaining tumor cells.

PURPOSE: This randomized phase II trial is studying surgery and thalidomide to see how well they work compared to surgery alone in treating patients with recurrent or metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the disease-free survival probability in patients with previously resected recurrent or metastatic colorectal carcinoma treated with adjuvant thalidomide vs placebo.
* Compare the time to recurrence in patients treated with these regimens.
* Determine whether serum/plasma levels of vascular endothelial growth factor and basic fibroblast growth factor preresection and postresection correlate with tumor recurrence and determine if these levels, as well as carcinoembryonic antigen (CEA) measurements, aid in predicting time to recurrence in these patients.
* Determine the pharmacokinetics and toxicity of long-term thalidomide therapy in these patients.
* Determine whether patients receiving thalidomide develop measurable antiangiogenic activity.
* Measure the presence of circulating tumor cells preresection and postresection and determine if this type of analysis can be used to predict recurrence in this patient population.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are stratified according to site of most recent lesion resection that rendered no evidence of disease (lung vs liver with no more than 3 lesions vs liver with more than 3 lesions vs lung and liver vs all other sites[including sites that were both resected and ablated]). Patients without evidence of residual disease are randomized to one of two treatment arms.

* Arm I: Patients receive oral thalidomide once daily.
* Arm II: Patients receive an oral placebo once daily. Treatment continues in both arms for 2 years in the absence of unacceptable toxicity or disease progression.

Patients are followed every 3 months for up to 3 years.

PROJECTED ACCRUAL: A total of 94 patients (47 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of recurrent or metastatic colorectal carcinoma previously resected within 12 weeks of study entry

  * Surgical resection combined with radiofrequency ablation allowed

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Hemoglobin at least 8.0 g/dL
* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Partial thromboplastin time (PTT)/prothrombin time (PT) no greater than 120% of control (except in therapeutically anticoagulated nonrelated medical conditions [e.g., atrial fibrillation])
* Total bilirubin no greater than 2.0 mg/dL (direct bilirubin no greater than 1.0 mg/dL for patients with Gilbert's syndrome)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) less than 2.5 times normal
* No history of hepatic cirrhosis
* No concurrent hepatic dysfunction

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No severe congestive heart failure or active ischemic heart disease
* No active clots within 1 year before diagnosis OR must be receiving concurrent treatment with anticoagulant (e.g., low molecular weight heparin or equivalent agent)

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 1 highly effective method of contraception AND 1 additional effective method of contraception for least 4 weeks before, during, and for at least 4 weeks after study participation
* No history of severe hypothyroidism
* No history of seizures
* No significant history of other medical problems that would preclude surgery
* No peripheral neuropathy greater than grade 1, except localized neuropathy due to a mechanical cause or trauma

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior biologic therapy

Chemotherapy:

* At least 4 weeks since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy

Surgery:

* See Disease Characteristics

Other:

* See Cardiovascular
* No concurrent sedating drugs that cannot be reduced to a minimal level
* No concurrent sedating recreational drugs or alcohol
* No concurrent antiseizure medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 1999-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven K. Libutti, MD, Study Chair — NCI - Surgery Branch
Locations (6):
- United States (6):
  - Center for Cancer Care at Goshen Health System, Goshen, Indiana
  - Suburban Hospital Cancer Program, Bethesda, Maryland
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - UPMC Cancer Center at UPMC Presbyterian, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1 - Thalidomide Once Daily | Arm 2 - Placebo Once Daily
Started | 23 | 16
Completed | 23 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 - Thalidomide Once Daily | Arm 2 - Placebo Once Daily | Total
Number analyzed (Participants) | 23 | 16 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 7 | 19
  >=65 years | 11 | 9 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.89 (8.70) | 71.19 (11.76) | 67.47 (10.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 15 | 9 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 22 | 16 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 17 | 13 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
  Hispanic | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 23 | 16 | 39

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Description: Time to progression was measured from the on study date until the date of progression or last follow up. Progression was assessed by the Response Evaluation Criteria for Solid Tumors (RECIST).Progressive Disease (PD)is at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions
Time Frame: 62 months
Population: The analysis was not done because there were not enough subjects to do any of the statistical analyses.
Arm/Group | Arm 1 - Thalidomide Once Daily | Arm 2 - Placebo Once Daily
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm 1 - Thalidomide Once Daily | Arm 2 - Placebo Once Daily
Serious Adverse Events (participants affected / at risk) | 5/23 | 4/16
Other Adverse Events (participants affected / at risk) | 11/23 | 6/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 - Thalidomide Once Daily (N=23) | Arm 2 - Placebo Once Daily (N=16)
AST (Hepatobiliary disorders) | 1 (1) | 0 (0)
CVA/TIA (Vascular disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Urethral obstruction (non-FDA reportable) (Renal and urinary disorders) | 1 (1) | 0 (0)
Abdominal pain (General disorders) | 0 (0) | 1 (1)
Cardiac-ischemia/infarction (Cardiac disorders) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Possible pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Swelling of uvula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 - Thalidomide Once Daily (N=23) | Arm 2 - Placebo Once Daily (N=16)
Anxiety (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety/Depression (Nervous system disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (6) | 2 (2)
Depression (Nervous system disorders) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0)
Euphoria (Nervous system disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 8 (8) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Libido (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Libido/impotence (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Pelvic pain (General disorders) | 1 (1) | 1 (1)
Peripheral neuropathy (Nervous system disorders) | 6 (7) | 5 (5)
Sedation (Nervous system disorders) | 1 (1) | 0 (0)
Skin changes (Skin and subcutaneous tissue disorders) | 8 (8) | 2 (2)
Weight gain (General disorders) | 2 (2) | 2 (2)
Headaches (Nervous system disorders) | 0 (0) | 1 (1)
PTT (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No